CLINICAL TRIAL: NCT01987882
Title: Outcomes of Hip Interventions for Children With Cerebral Palsy - An International Multi-centre Prospective Comparative Cohort Study
Brief Title: Cerebral Palsy Hip Outcomes Project - International Multi-centre Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Other Study IDs: 313575
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
Keywords: Outcomes research, treatment effectiveness, quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- A. "Natural" History or Watchful Waiting
- B. Serial Botulinum Toxin Injections +/- Abduction Bracing
- C. Adductor (+/- psoas) Muscle Releases Alone
- D. Hip Reconstructive Surgery
- E. Salvage Hip Surgery

SUMMARY:
The primary purpose of the project is to evaluate the effectiveness of different intervention strategies to prevent or relieve symptoms associated with hip instability in children with severe cerebral palsy, using the validated Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD©) questionnaire as the primary outcome measure of health-related quality of life for this population.

DETAILED DESCRIPTION:
Background: Children with severe cerebral palsy (CP) are at high risk for dislocating their hips. These hips are associated with contractures and pain, which can interfere with care-giving, seating, positioning, mobility and quality of life. The primary purpose of this project (Aim 2) is to evaluate the effectiveness of different intervention strategies to prevent or relieve the symptoms associated with hip instability in children with severe non-ambulatory CP, using the validated Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD©) questionnaire as the primary outcome measure of health related quality of life (HRQL) for this population. Secondarily, this project will also measure the impact of hip displacement on HRQL of these children. This project will be the first of its kind and this scale, which will systematically study the impact of hip instability and its management in children with severe CP, using a meaningful outcome measure that was developed specifically for this purpose. The international network of investigators/sites and the infrastructure established for this project will facilitate the long term follow-up of the participants in this study, as well as the conduct of other multi-centre clinical trials and cohort studies to evaluate the effectiveness of current and future interventions aimed at improving the quality of life of children with severe disabilities.

Study Design & Participants: International multi-centre prospective longitudinal cohort study of children with severe (non-ambulant) cerebral palsy (GMFCS levels IV & V) from ages 3 to 18 who have radiographic evidence of hip displacement [Reimer's Migration Percentage (MP) ≥ 30%].

Measures: Detailed demographic information, and prognostic factors, including co-morbid conditions will be recorded at baseline, in addition to self-administered parental reports of HRQL as measured by the CPCHILD. Hip status will be classified using standardized radiographic measures of Reimer's MP and acetabular index (AI). The primary outcome measure CPCHILD, as well as the MP & AI will be measured at 6, 12 and 24 months following initial intervention.

Aim 1: Measure the impact of increasing hip displacement in children with severe (non-ambulant) CP on their HRQL as measured by the CPCHILD questionnaire.

Aim 2: (Primary Purpose): Measure the effectiveness of different strategies of interventions for hip displacement in children with severe (non-ambulant) CP in a prospective longitudinal comparative cohort study using the CPCHILD as the primary outcome measure of HRQL.

Aim 3: Compare the types and rates of adverse events and complications associated with each of the treatment cohorts.

Methods: Observational study of usual (site/surgeon specific) clinical practice. Investigators at each site will enroll eligible participants and assign each to one of the following 5 cohorts based on individual treating doctor's &/or parental preferences:

A. "Natural" history or watchful waiting (N=100)

B. Serial botulinum toxin injections +/- abduction bracing (N=100)

C. Adductor (+/- psoas) muscle releases alone (N=100)

D. Hip reconstructive surgery (N=100)

E. Salvage hip surgery (N=100)

The baseline MP and CPCHILD scores for all participants will be analyzed cross-sectionally to evaluate the correlation between hip displacement and the CPCHILD scores to serve Aim 1. For Aim 2, children undergoing interventions for hip instability (Groups B, C, D, & E) will be compared with each other as well as with their respective matched counterparts of untreated children (Group A), using repeated measures of analysis of covariance (ANOCOVA) to measure the mean change in scores from baseline at 6, 12 and 24 months after intervention.

Timelines: 500 participants will be recruited in 24 months, and followed for 24 months. The analysis, reporting of results, manuscript development and knowledge transfer will take 12 months. In total, the study will take 5 years to complete.

ELIGIBILITY:
Inclusion Criteria:

* Children with a working diagnosis of cerebral palsy or cerebral palsy-like condition
* Between 2 to 18 years of age
* Has a migration percentage ≥ 30%
* Non-ambulatory; the primary mode of mobility is a wheelchair
* Parent/primary caregiver must understand one of the languages in which the CPCHILD has been translated, culturally adapted and validated.

Exclusion Criteria:

* History of prior hip surgery
* Received botulinum toxin injection within the previous 3 months. Recruitment will be delayed until at least 3 months after prior botulinum toxin injection.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with severe, non-ambulant cerebral palsy (GMFCS level IV and V) and their parent / primary caregiver will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-06; Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
CPCHILD questionnaire: Total Score (0-100) | Change from baseline to 12 months after treatment
  The primary outcome measure will be based at the 12 month assessment. The CPCHILD questionnaire is a validated outcome measure of health-related quality of life specifically developed for children with severe, non-ambulant cerebral palsy (GMFCS level IV and V) to evaluate the effectiveness of different treatment options.

SECONDARY OUTCOMES:
CPCHILD Questionnaire: Total Score (0-100) | Change from baseline to 24 months after treatment
  The CPCHILD questionnaire is a validated outcome measure of health-related quality of life specifically developed for children with severe, non-ambulant cerebral palsy (GMFCS level IV and V) to evaluate the effectiveness of different treatment options.
Reimer's Migration Percentage (MP) | Change from baseline to 24 months after treatment
  The Reimer's Migration Percentage (MP) quantifies the magnitude of the displacement of the femoral head that is uncovered by the acetabulum.
Acetabular Index (AI) in degrees | Change from baseline to 24 months after treatment
  The Acetabular Index (AI) in degrees quantifies the magnitude of acetabular dysplasia.
Morphological Hip Classification in Cerebral Palsy (MHC) | Change from baseline to 24 months after treatment
  The Morphological Hip Classification in Cerebral Palsy (MHC) describes the sphericity of the femoral head.
CPCHILD Questionnaire: Subscale Scores (0 - 100) | Change from baseline to 24 months after treatment
  The Subscale scores of the CPCHILD© questionnaire represent the following domains:
  1. Activities of Daily Living/Personal Care (9 items);
  2. Positioning, Transferring & Mobility (8);
  3. Comfort & Emotions (9);
  4. Communication & Social Interaction (7);
  5. Health (3);
  6. Overall Quality of Life (1).
  Standardized scores are generated on a scale of 0 (worst) to 100 (best) for each of the 6 domains.

OTHER OUTCOMES:
Adverse Events and Complications | Adverse events will be recorded up to 24 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Unni Narayanan, MBBS, MSc, FRCSC, Principal Investigator — Holland Bloorview Kids Rehab and The Hospital for Sick Children, Toronto, Canada
Locations (27):
- United States (9):
  - Shriners Hospitals for Children - Northern California, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Children's Hospital Boston, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Children's of Mississippi, Jackson, Mississippi
  - Hospital for Special Surgery, New York, New York
  - New York-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Royal Children's Hospital, Melbourne, Victoria, Australia
- Canada (4):
  - BC Children's Hospital, Vancouver, British Columbia
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Shriners Hospital for Children - Canada, Montreal, Quebec
- Aarhus University Hospital, Aarhus, Denmark
- Safra Hospital for Children, Tel Litwinsky, Ramat Gan, Israel
- Starship Children's Hospital of New Zealand, Auckland, New Zealand
- K. Marcinkowski Medical University, Poznan, Poland
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea
- Sweden (2):
  - Lund University Hospital, Lund
  - Astrid Lindgren's Children's Hospital, Stockholm
- United Kingdom (6):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry, England
  - Alder Hey Children's NHS Foundation Trust, Liverpool, England
  - Royal National Orthopaedic Hospital, London, England
  - The Royal London and St. Bartholomew's Hospitals, London, England
  - Nuffield Orthopaedic Centre NHS Trust, Oxford, England
  - Royal Hospital for Sick Children, Edinburgh, Scotland

REFERENCES:
- [Background] Narayanan UG, Fehlings D, Weir S, Knights S, Kiran S, Campbell K. Initial development and validation of the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD). Dev Med Child Neurol. 2006 Oct;48(10):804-12. doi: 10.1017/S0012162206001745. PMID 16978459
- [Derived] Miller SD, Juricic M, Fajardo N, So J, Shore BJ, Narayanan UG, Mulpuri K. Variability in Postoperative Immobilization and Rehabilitation Following Reconstructive Hip Surgery in Nonambulatory Children With Cerebral Palsy. J Pediatr Orthop. 2021 Aug 1;41(7):e563-e569. doi: 10.1097/BPO.0000000000001850. PMID 33999564
- See also: Website of the CPCHILD© Project — http://www.sickkids.ca/Research/CPCHILD-Questionaire/CPCHILD-Project/index.html